CLINICAL TRIAL: NCT06725914
Title: The Effect of Kangaroo Father Care Transport on Physiological Parameters, Anxiety and Paternal Attachment in Preterm Infants: A Randomized Controlled Study
Brief Title: The Effect of Kangaroo Father Care Transport on Preterm Infants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Büşra GÜÇLÜ (Other)
Collaborators: Selcuk University (Other)
Responsible Party: Sponsor-Investigator, Zeynep Büşra GÜÇLÜ, Nurse, Selcuk University
Organization: Selcuk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Selcuk University Health Care
Record Dates: First submitted 2024-11-26; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Nurse's Role; Preterm Birth; Fathers
Keywords: Father; Early kangaroo care; preterm infant; nurse; transport
MeSH Terms: conditions — Premature Birth | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Intervention Model Description: The study was a single-blind, parallel group, randomized controlled experimental design.Randomization was performed by an independent investigator to avoid bias. Preterm infants were randomly assigned to the experimental and control groups (1:1) by simple randomization method. Using the permutation block randomization method, 6 permutations were formed as a block of 4 using the letters A and B. The number of samples was divided by the number of permutations (40/6=7) and sorted 7 times from 1 to 6 using a table of random numbers (www.randomizer.org). The combinations generated according to this order (e.g. BBAA (3) ABBA (2)) were prepared in sealed envelopes (40 pieces) by an independent statistician. Which letter represented which group was determined by lottery. To ensure confidentiality, each preterm infant was randomly assigned a numerical code and the results were reported to the researcher collectively in sealed opaque envelopes.
Who Masked: Outcomes Assessor
Masking Description: In this study, statistician blinding was used for the implementation of randomization and data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation of paternal early kangaroo care transport (Experimental): Early kangaroo care was administered immediately after delivery. The fathers were seated on a wheelchair for transportation from the gynecology operating room to the NICU. The newborn was then dressed in a diaper and hat. The preterm baby was laid naked on the father's bare chest in an upright position. Preterms were secured with a kangaroo care garment in the frog leg position in the prone position with the head turned to the side. The baby was covered with a blanket to prevent heat loss.
  Interventions: Behavioral: kangaroo care
- Control Group (No Intervention): The babies in the control group were transported to the NICU in the arms of the nurse after birth as in the clinical routine.

INTERVENTIONS:
Behavioral: kangaroo care — Transport practice with paternal kangaroo care in preterm infants
  Arms: Implementation of paternal early kangaroo care transport

SUMMARY:
This study was planned to investigate the effect of paternal kangaroo care and transport on physiologic parameters, anxiety and paternal attachment in preterm infants.

DETAILED DESCRIPTION:
This study was conducted to determine the effects of paternal kangaroo care and transport of preterm infants on the physiologic parameters of the infant and the anxiety and attachment levels of the fathers.

ELIGIBILITY:
Inclusion Criteria:Neonatal related;

* Born by caesarean section,
* Born at 34-36+6 weeks gestation,
* Apgar score of 7 and above at 1 and 5 minutes,
* Stable and healthy,
* Infants with a body weight of 1500 g and above were included. It's about the father;
* Who volunteered to participate in the study,
* No mental and psychological problems,
* No communication problems (speech, hearing and severe visual impairment),
* Fathers who did not carry contact-transmitted diseases (Covid-19, herpes simplex, scabies, etc.) were included.

Exclusion Criteria:- Congenital anomalies,

* Abdominal defects such as ompholocele, diaphragmatic hernia, gastroschisis,
* Receiving invasive and noninvasive respiratory support,
* With chest tube and umbilical catheter,
* Foreign babies and their fathers were ostracized.

Ages: 34 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-12-03 (Actual); Primary Completion 2024-06-16 (Actual); Study Completion 2024-12-24 (Estimated)

PRIMARY OUTCOMES:
Physiological Parameter Monitoring Form-Heart Rate | 3 minutes before the intervention
  Heart Rate in the Physiologic Parameter Monitoring Form was measured 3 minutes before (T0) the intervention.
Physiological Parameter Monitoring Form-SPO2 | 3 minutes before the intervention
  SPO2 in the Physiologic Parameter Monitoring Form was measured 3 minutes before (T0) the intervention.
Physiological Parameter Monitoring Form-Body temperature (°C) | 3 minutes before the intervention
  Body temperature (°C) in the Physiologic Parameter Monitoring Form was measured 3 minutes before (T0) the intervention.
Father-Infant Information Form-Paternal characteristics, maternal characteristics and infant characteristics | 15 minutes before the intervention
  Paternal characteristics (age, number of children, educational status, employment status, income status and kangaroo care experience), maternal characteristics (age, educational status, employment status, health problems during pregnancy) and infant characteristics (date of birth, gestational week, gender, birth weight, birth length, birth head circumference, APGAR score, type of anesthesia at birth) were recorded before the intervention.
State Anxiety Scale | 15 minutes before the intervention
  State Anxiety Scale was recorded 15 minutes before the intervention.
Father-Infant Attachment Scale | 15 minutes before the intervention
  Father-Infant Attachment Scale was recorded 15 minutes before the intervention.

SECONDARY OUTCOMES:
Physiological Parameter Monitoring Form-Heart Rate | 3 minutes after the end of kangaroo care (T2).
  Heart Rate in the Physiologic Parameter Monitoring Form was measured 3 minutes after (T2) the end of kangaroo care
Physiological Parameter Monitoring Form-Heart Rate | 3 minutes after initiation of transport with kangaroo care.(T1)
  Heart Rate in the Physiologic Parameter Monitoring Form was measured 3 minutes after (T1) initiation of transport with kangaroo care.
Physiological Parameter Monitoring Form-SPO2 | 3 minutes after initiation of transport with kangaroo care.(T1)
  SPO2 in the Physiologic Parameter Monitoring Form was measured 3 minutes after (T1) initiation of transport with kangaroo care.
Fizyolojik Parametre İzleme Formu-SPO2 | 3 minutes after the end of kangaroo care (T2)
  SPO2 in the Physiologic Parameter Monitoring Form was measured 3 minutes after (T2) the end of kangaroo care
Physiological Parameter Monitoring Form-Body temperature (℃) | 3 minutes after initiation of transport with kangaroo care.(T1)
  Body temperature (℃) in the Physiologic Parameter Monitoring Form was measured 3 minutes after (T1) initiation of transport with kangaroo care.
Physiological Parameter Monitoring Form-Body temparature (℃) | 3 minutes after the end of kangaroo care (T2).
  Body temparature (℃) in the Physiologic Parameter Monitoring Form was measured 3 minutes after (T2) the end of kangaroo care
State Anxiety Scale | 15 minutes before the intervention (T2)
  State Anxiety Scale 15 minutes after the end of the intervention (T2)
Father-Infant Attachment Scale | 15 minutes after the intervention.
  Father-Infant Attachment Scale was recorded 15 minutes after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- SELÇUK University, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Background] Yildirim F, Buyukkayaci Duman N, Sahin E, Vural G. The Effect of Kangaroo Care on Paternal Attachment: A Randomized Controlled Study. Adv Neonatal Care. 2023 Dec 1;23(6):596-601. doi: 10.1097/ANC.0000000000001100. Epub 2023 Oct 26. PMID 37884013
- [Background] Unal Toprak F, Senturk Erenel A. Impact of kangaroo care after caesarean section on paternal-infant attachment and involvement at 12 months: A longitudinal study in Turkey. Health Soc Care Community. 2021 Sep;29(5):1502-1510. doi: 10.1111/hsc.13210. Epub 2020 Oct 28. PMID 33118268
- [Background] Varela N, Tessier R, Tarabulsy G, Pierce T. Cortisol and blood pressure levels decreased in fathers during the first hour of skin-to-skin contact with their premature babies. Acta Paediatr. 2018 Apr;107(4):628-632. doi: 10.1111/apa.14184. Epub 2017 Dec 29. PMID 29224247
- [Background] Bodet LM, Danielo M, Roze JC, Flamant C, Muller JB. Father newborn skin-to-skin wheelchair transfer from delivery room to neonatal care unit: Possible change in practices. Arch Pediatr. 2022 Feb;29(2):100-104. doi: 10.1016/j.arcped.2021.11.005. Epub 2022 Jan 14. PMID 35039187
- [Background] Pujara RK, Upadhyay V, Thacker JP, Rana BB, Patel SS, Joshi JM, Shinde MK, Nimbalkar SM, Patel DV. Efficacy of skin-to-skin vs. cloth-to-cloth contact for thermoregulation in low birth weight newborns: a randomized crossover trial. J Trop Pediatr. 2023 Feb 6;69(2):fmad013. doi: 10.1093/tropej/fmad013. PMID 36811579
- [Background] Cristobal Canadas D, Bonillo Perales A, Galera Martinez R, Casado-Belmonte MDP, Parron Carreno T. Effects of Kangaroo Mother Care in the NICU on the Physiological Stress Parameters of Premature Infants: A Meta-Analysis of RCTs. Int J Environ Res Public Health. 2022 Jan 5;19(1):583. doi: 10.3390/ijerph19010583. PMID 35010848
- [Background] Tas Arslan F, Akkoyun S, Kucukoglu S, Kocoglu-Tanyer D, Konak M, Soylu H. Effect of kangaroo mother care on cerebral oxygenation, physiological parameters, and comfort levels in late-premature infants: A randomized controlled trial. Midwifery. 2024 Oct;137:104096. doi: 10.1016/j.midw.2024.104096. Epub 2024 Jul 7. PMID 39024964
- [Background] Durmaz A, Sezici E, Akkaya DD. The effect of kangaroo mother care or skin-to-skin contact on infant vital signs: A systematic review and meta-analysis. Midwifery. 2023 Oct;125:103771. doi: 10.1016/j.midw.2023.103771. Epub 2023 Jul 10. PMID 37454580